CLINICAL TRIAL: NCT01972945
Title: Vaginoscopy Against Standard Treatment (VAST): a Randomised Controlled Trial
Acronym: VAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Thomas Justin Clark, Consultant Obstetrician and Gynaecologist, Birmingham Women's NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VAST
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Hysteroscopy Technique
Keywords: vaginoscopy; hysteroscopy; office hysteroscopy; outpatient hysteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginoscopy (Experimental): Vaginoscopy, otherwise known as the 'no touch' technique, describes a technique where the hysteroscope is guided into the uterus without the need for potentially painful vaginal instrumentation i.e. passage of a vaginal speculum to separate the vaginal walls, cleansing of the cervix and sometimes application of traumatic forceps to the ectocervix in order to stabilise it.
  Interventions: Procedure: Vaginoscopy
- Standard Hysteroscopy (Active Comparator): Traditional hysteroscopy consists of introducing speculum and grasping of the cervix to provide counter traction to allow instrumentation of the uterus. Introducing a speculum also allows the cervix to be cleaned with sterilising fluid.
  Interventions: Procedure: Standard Hysteroscopy

INTERVENTIONS:
Procedure: Vaginoscopy — Vaginoscopy, otherwise known as the 'no touch' technique, describes a technique where the hysteroscope is guided into the uterus without the need for potentially painful vaginal instrumentation i.e. passage of a vaginal speculum to separate the vaginal walls, cleansing of the cervix and sometimes application of traumatic forceps to the ectocervix in order to stabilise it.
  Other Names: no touch technique
  Arms: Vaginoscopy
Procedure: Standard Hysteroscopy — Traditional hysteroscopy consists of introducing speculum and grasping of the cervix to provide counter traction to allow instrumentation of the uterus. Introducing a speculum also allows the cervix to be cleaned with sterilising fluid.
  Arms: Standard Hysteroscopy

SUMMARY:
Inserting a telescope into the womb to identify and treat problems with bleeding, pain or reproduction is the commonest surgical intervention in gynaecology. This procedure is known as a 'hysteroscopy'. The established 'traditional' technique for introducing the hysteroscope into the womb involves the use of a 'speculum', which is inserted into the vagina. A speculum is the metal or plastic instrument used to stretch and separate the vaginal walls so that the opening to the womb, known as the 'cervix' can be seen. The cervix is then cleaned and frequently grasped with a sharp toothed forcep to provide traction before the hysteroscope is inserted. Whilst hysteroscopy is safe, it is known that pain during the procedure can lead to a poor patient experience, and even trigger fainting episodes or failure to complete the procedure. As the hysteroscopes have become smaller, it has been recognised that it is possible to access the cervix and womb (i.e. 'uterus') directly using the hysteroscopic vision without inserting any of these potentially pain inducing vaginal instruments. There is however, uncertainty whether this newer technique known as 'vaginoscopy' or the 'no touch technique' will minimise the pain experienced by the patient or reduce the propensity to fainting. Futhermore, even if vaginoscopy is shown to be less painful, the technique may be more prone to failure due to an inability to transverse the cervix and enter the uterus without additional instruments. Post-operative infection rates of the uterus may also be higher due to vaginal contamination.

Reducing pain and complications and improving success of the procedure as well as optimising patients experience is important because hysteroscopy is an intimate examination, known to be associated with significant anxiety and pain. Furthermore, the procedure is widely practised representing the most common surgical intervention in day-to-day gynaecological practice in the UK and elsewhere. It is therefore important, and timely given that outpatient hysteroscopy is increasing especially in community settings, that a large, high quality randomised controlled trial comparing 'vaginoscopy' and the 'traditional' hysteroscopy is undertaken to resolve the uncertainty as to whether vaginoscopy is less painful, safe and more successful than existing approaches to hysteroscopy.

DETAILED DESCRIPTION:
1. Background

   Office hysteroscopy can be associated with significant anxiety, pain and patient dissatisfaction (Clark et al.). One technical modification identified to potentially reduce pain at hysteroscopy is 'vaginoscopy', otherwise known as the 'no touch' technique (Busquets and Lemus, 1993; Clark and Gupta, 2005; Cooper et al., 2010). This describes a technique where the hysteroscope is guided into the uterus without the need for potentially painful vaginal instrumentation. Pain is often experienced by the patient at a number of stages during the standard hysteroscopy practice, these include passage of a vaginal speculum to separate the vaginal walls in order to visualise the cervix, cleansing of the cervix and sometimes application of traumatic forceps to the ectocervix in order to stabilise it. Vaginoscopy could be less traumatic because the approach minimises potentially painful manoeuvres in the lower genital tract.

   Recent technological advances have led to the miniaturisation of hysteroscopes, which facilitates vaginoscopy by reducing resistance to advancement of the hysteroscope through the relatively narrow and often tortuous cervical canal. However, despite these modifications in instrumentation, few clinicians use vaginoscopy routinely preferring more invasive traditional approaches. This may reflect a lack of familiarity with the technique as well as concerns over the ability to identify and traverse the cervical canal in order to access the uterine cavity.

   We therefore designed a randomised controlled trial (RCT) to compare standard approach to hysteroscopy against vaginoscopy evaluating important clinical outcomes such as pain, feasibility, acceptability, vasovagal responses and infection. To inform the study design we conducted pilot work including a survey of gynaecological endoscopists, and a systematic review of the current evidence.
2. Systematic review and meta-analysis

   We have previously completed and reported a systematic review and meta-analysis of vaginoscopy compared to standard hysteroscopy (Cooper et al., 2010). The databases searched included MEDLINE, EMBASE, and CINAHL using a combination of the keyword 'hysteroscopy', 'vaginoscopy', vaginoscop*', 'no-touch', and their associated word variants and medical subject headings. The Cochrane Library was searched using the keywords 'hysteroscopy', 'vaginoscopy', 'vaginoscopic' and 'no-touch'.

   Of the 1167 citations retrieved, six studies met the criteria for inclusion and in four there was suitable data for meta-analysis. Vaginoscopy was found to be less painful than traditional approaches, with a standard mean difference in visual analogue scales (VAS) pain scores of -0.44 (95% CI -0.65 to -0.22)(Cooper et al., 2010). However there was statistically significant heterogeneity and this was also seen in the wide variation in procedure feasibility (failure rates varying from 2% to 17%) (Cooper et al., 2010). This inconsistency reflected the lack of standardisation of approach both in relation to vaginoscopy and traditional speculum based approaches where there was variation between studies in the administration of local cervical anaesthesia, application of cervical tenaculum forceps, and the size and angle of the rigid hysteroscope employed. None of these small RCTs (Almeida et al., 2008; Garbin et al., 2006; Guida et al., 2006; Paschopoulos et al., 1997; Sagiv et al., 2006; Sharma et al., 2005) had optimal randomisation processes in terms of using computer generated random number sequences and third party concealment. The review and subsequent Royal College of Obstetrics and Gynaecology (RCOG) guideline (Clark et al.; Cooper et al., 2010) recommended further higher quality adequately powered RCTs to examine more comprehensively the role of vaginoscopy in terms of pain, feasibility, acceptability and complications.
3. The need for a RCT comparing vaginoscopy to standard hysteroscopy

   The current restricted use of vaginoscopy is likely to be the result of a lack of experience with the technique and uncertainty as to whether the technique is associated with a worthwhile reduction in procedural pain and improvement in patient acceptability. Furthermore, there is concern that vaginoscopy is technically more challenging leading to prolonged procedures which may fail to be completed, lead to more vaso-vagal fainting episodes and a higher likelihood of post-operative infection of the uterus.

   In view of the uncertainty over the effectiveness of vaginoscopy we designed an RCT. The aim was to evaluate whether vaginoscopy or standard hysteroscopy was potentially more successful in the office setting by comparing failure rates, complications, infection rates, patient acceptability, and pain scores. In the first instance we designed a feasibility pilot trial (VAginoscopy versus Standard Teloscope for office hysteroscopy trial; VAST) to inform the design, conduct and feasibility of a larger scale RCT.
4. Objectives

   1. To estimate whether the vaginoscopic technique is potentially more successful compared to traditional approaches where success is defined as a completed diagnostic hysteroscopy with an acceptable level of patient reported pain without a vasovagal episode or post-operative uterine infection.
   2. To test the hypothesis that the success of vaginoscopy differs according to parity, menopausal status, obesity and cervical surgery.
   3. To test the hypothesis that in women undergoing an office hysteroscopy, a vaginoscopic technique is associated with on average at least 10% less pain (as measured by visual analogues scores) compared to traditional approaches.
   4. To test the hypothesis that in women undergoing an office hysterosocpy, a vaginoscopic technique is associated with fewer vaso-vagal episodes compared to traditional approaches.
   5. To test the hypothesis that in women undergoing an office hysteroscopy, there is no difference in the rates of failure to complete the procedure between vaginoscopy and traditional approaches.
   6. To test the hypothesis that in women undergoing an office hysteroscopy, there is no difference in the incidence of post-operative uterine infection between vaginoscopy and traditional approaches.
   7. To test the hypothesis that in women undergoing an office hysteroscopy, a vaginoscopic technique is associated with better patient acceptability.
5. References

Almeida, Z.M.M.C. de, Pontes, R., and Costa, H. de L.F.F. (2008). [Evaluation of pain in diagnostic hysteroscopy by vaginoscopy using normal saline at body temperature as distension medium: a randomized controlled trial]. Rev. Bras.

Ginecol. E Obstetrícia Rev. Fed. Bras. Soc. Ginecol. E Obstetrícia 30, 25-30.

Busquets, M., and Lemus, M. (1993). [Practicability of panoramic hysteroscopy with CO2. Clinical experience: 923 cases]. Rev. Chil. Obstet. Ginecol. 58, 113-118.

Clark, T.J., and Gupta, J.K. (2005). Handbook of outpatient hysteroscopy: a complete guide to diagnosis and therapy (CRC Press).

Clark, T.J., Cooper, N.A., and Kremer, C. Best practice in outpatient hysteroscopy.

Cooper, N.A.M., Smith, P., Khan, K.S., and Clark, T.J. (2010). Vaginoscopic approach to outpatient hysteroscopy: a systematic review of the effect on pain. BJOG Int. J. Obstet. Gynaecol. 117, 532-539.

Garbin, O., Kutnahorsky, R., Göllner, J.L., and Vayssiere, C. (2006). Vaginoscopic versus conventional approaches to outpatient diagnostic hysteroscopy: a two-centre randomized prospective study. Hum. Reprod. Oxf. Engl. 21, 2996-3000.

Guida, M., Di Spiezio Sardo, A., Acunzo, G., Sparice, S., Bramante, S., Piccoli, R., Bifulco, G., Cirillo, D., Pellicano, M., and Nappi, C. (2006). Vaginoscopic versus traditional office hysteroscopy: a randomized controlled study. Hum. Reprod. Oxf. Engl. 21, 3253-3257.

Paschopoulos, M., Paraskevaidis, E., Stefanidis, K., Kofinas, G., and Lolis, D. (1997). Vaginoscopic approach to outpatient hysteroscopy. J. Am. Assoc. Gynecol. Laparosc. 4, 465-467.

Sagiv, R., Sadan, O., Boaz, M., Dishi, M., Schechter, E., and Golan, A. (2006). A new approach to office hysteroscopy compared with traditional hysteroscopy: a randomized controlled trial. Obstet. Gynecol. 108, 387-392.

Sharma, M., Taylor, A., di Spiezio Sardo, A., Buck, L., Mastrogamvrakis, G., Kosmas, I., Tsirkas, P., and Magos, A. (2005). Outpatient hysteroscopy: traditional versus the "no-touch" technique. BJOG Int. J. Obstet. Gynaecol. 112, 963-967.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16years or over
* Referred for diagnostic of operative hysteroscopy in the outpatient setting
* Written informed consent obtained prior to the hysteroscopy

Exclusion Criteria:

* Need for hysteroscopic surgical intervention that requires cervical dilatation e.g. Novasure uterine ablation

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Hysteroscopy success (composite primary outcome) | At the time of surgery (day 1) for all elements except for infection (day 14)
  The primary clinical outcome is a composite outcome of a completed hysteroscopy with an acceptable level of patient reported pain without a vasovagal episode or post-operative uterine infection. A composite outcome has been chosen as it was felt that all of these factors are important to classify a hysteroscopy as successful. See individual elements in secondary outcomes for a description of how they will be measured

SECONDARY OUTCOMES:
Procedure Pain | At the time of surgery (day 1)
  The main limitation of outpatient interventions is the amount of pain generated. Visual analogue scales (VAS) originally devised as measured of well-being have been successfully adapted to measure pain. This technique involves use of 10cm line of a piece of paper representing a continuum of the patients' opinion of the degree of pain. It is explained to the patient that the one extreme of the line represent "no pain at all" while the other represents "as much pain as she can possibly imagine". The subject rates the degree of pain by placing a mark on the line and scale values are obtained by measuring the distance from zero to that mark. The reliability of visual analogue scales in the assessment of pain has established as reproducible and accurate. A baseline pain questionnaire will be administered before the procedure and a further pain assessment will be made immediately after treatment.
Procedure failures | At the time of surgery (day 1)
  Part of the primary clinical outcome is to test whether the vaginoscopic technique reduces the number of procedure failures. Unfortunately, it is occasionally necessary to abandon outpatient hysteroscopic procedure normally because of pain or anxiety. The clinician will collect this data on the treatment form.
Infection rates | Two weeks post procedure (day 14)
  The patient will be contacted two weeks after the procedure. An infection will be defined as any of the following in the two-week period after the procedure:
  1. If the patient has received antibiotics for a urinary tract infection
  2. If the patient has received antibiotics for vaginal discharge
  3. If the patient reports 2 out of the following 3 symptoms: offensive vaginal discharge, pelvic pain and pyrexia.
Vasovagal episodes | At the time of surgery (day 1)
  Another part of the primary outcome is assessing whether vaginoscopy reduces the number of vasovagal episodes. Vaso-vagal reactions will be defined clinically as patient is unable to leave operating couch within 5minutes of cessation of procedure due to feeling faint or dizzy or nauseous. The clinical will collect this data on the treatment form.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Clark, MD(hons), Principal Investigator — Birmingham Women's NHS Foundation Trust
Locations (1):
- Birmingham Womens Hospital, Birmingham, West Midlands, United Kingdom